CLINICAL TRIAL: NCT06596317
Title: Impact of Indigo Carmine Pump Spraying on the Adenoma Detection Rate: A Randomized Controlled Trial
Brief Title: Impact of Indigo Carmine Pump Spraying on the Adenoma Detection Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022SDU-QILU-294
Record Dates: First submitted 2023-04-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyps; Adenomatous Polyps; Adenoma Detection Rate; Chromoendoscopy; Colorectal Neoplasms
Keywords: Adenoma Detection Rate; Chromoendoscopy; Colonoscopy; Colorectal Cancer; Indigo Carmine; Mean Adenoma Per Patient
MeSH Terms: conditions — Colonic Polyps; Adenomatous Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chromoendoscopy with indigo carmine solution spray (Experimental): Patients in this group will be carefully observed with spraying indigo carmine solution during the colonoscopy withdraw.
  Interventions: Procedure: Chromoendoscopy
- Conventional colonoscopy without indigo carmine solution spray (Active Comparator): Patients in this group will be carefully observed without spraying anything during the colonoscopy withdraw.
  Interventions: Procedure: Conventional colonoscopy

INTERVENTIONS:
Procedure: Chromoendoscopy — Patients will undergo chromoendoscopy with spraying indigo carmine.
  Arms: Chromoendoscopy with indigo carmine solution spray
Procedure: Conventional colonoscopy — Patients will undergo conventional colonoscopy.
  Arms: Conventional colonoscopy without indigo carmine solution spray

SUMMARY:
Detection and removal of polyps during colonoscopy is crucial for the prevention of colorectal cancer. Indigo carmine spraying up to the colonic mucosa could probably increase the adenoma detection rate. The traditional method of dye spraying with spraying catheter or syringe would consume a lot of time and dye volume. Now, the more convenient auxiliary water supply channel can be used to spray indigo carmine. In order to explore the clinical application value of spraying indigo carmine solution by auxiliary water channel in high-risk population, we performed a prospective, randomized controlled trial to compare adenoma detection rate of conventional colonoscopy and chromoendoscopy.

DETAILED DESCRIPTION:
If patients scheduled for colonoscopy meet the inclusion criteria but not the exclusion criteria, he or she will be recruited to the study and randomized to one of two groups. Subjects in Group A (treatment group) will undergo colonoscopy with spraying indigo carmine solution during withdrawal process. Subjects in Group B (control group) will undergo a standard conventional colonoscopy without spraying any solution during withdrawal process. The traditional method of dye spraying with spraying catheter or syringe would consume a lot of time and dye volume. The solution spraying process was implemented by a water jet channel using auxiliary foot pump. Any lesions found during the procedure will be removed and sent for pathological examination. The investigator will record the patient's general information (such as gender, age, symptoms, body mass index， etc.), colonoscopy data (such as duration, dye amount, etc.), and lesion characteristics (such as location, morphology, histopathological classification, etc.). Randomization was done with SPSS program. All data were analyzed according to the ITT analysis, and the PP analysis was performed for all outcomes. Continuous variables were presented as means ± standard deviation (SD), and compared using the Student t test. Categorical data were expressed as number with percentage and analyzed using the chi-squared test or the Fisher exact test. All statistical analyses were performed using IBM SPSS Statistics or R Statistics, and 2-sided P<0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of colorectal cancer or colorectal adenoma
* Patients whose first-degree relatives have a history of colorectal cancer or colorectal adenoma
* Patients with gastrointestinal symptoms (abdominal pain, bloody stool, chronic diarrhea or constipation, Unexplained anemia or weight loss;
* Patients with positive fecal occult blood tests

Exclusion Criteria:

* Patients with severe comorbidity
* Patients who are not suitable for colonoscopy
* Patients who received urgent or therapeutic colonoscopy
* Patients with pregnancy, inflammatory bowel disease, polyposis syndromes, suspected CRC; intestinal obstruction, coagulopathy
* Patients with aspirin, clopidogrel or other anticoagulants/ antiplatelet drugs intake within 7 days
* Patients with failed cecal intubation
* Patients with inadequate bowel preparation quality (Boston score ≤5)
* Patients who refuse to participate or to provide informed consent

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate(ADR) | procedure time
  ADR was calculated as the number of patients with at least one adenoma divided by the total number of patients. In other words, the adenoma detection rate of the sample was the proportion of patients with adenoma detected.

SECONDARY OUTCOMES:
detected rate of different lesions | procedure time
  Lesions are classified according to their size, location, morphology and histopathology, the corresponding detection rate was calculated as secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Ji, MD, PHD, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China